CLINICAL TRIAL: NCT02359006
Title: The Effects of Minocycline on Opioid-induced Hyperalgesia in Opioid-Maintained Patients
Brief Title: The Effects of Minocycline in Opioid-maintained Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1412015119; 2T32DA007238-26 (NIH)
Record Dates: First submitted 2015-02-03; First posted 2015-02-09 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Opioid Dependence; Pain
Keywords: Analgesia; pain analgesia; methadone; opiates
MeSH Terms: conditions — Opioid-Related Disorders; Pain; Agnosia | interventions — Minocycline; Tetracycline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- minocycline (Active Comparator): 200mg minocycline
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — Minocycline will be compared with placebo
  Other Names: tetracycline
  Arms: minocycline
Drug: Placebo — Placebo will be compared with minocycline
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Opioids are the most commonly utilized pharmacological treatment for moderate to severe pain. However, their clinical value is hindered by the development of opioid-induced hyperalgesia (OIH). OIH manifests as heightened pain sensitivity, and is an increasingly challenging drawback to the efficacy of opioid treatment. Although the mechanism of action modulating OIH is not completely understood, previous animal studies suggest that this phenomenon is a result of proinflammatory responses. Thus, administering an adjunct anti-inflammatory agent may attenuate OIH. Minocycline is one such agent; it is a tetracycline derivative antibiotic that inhibits microglia activation, nitric oxide (NO) production, and the release of pro-inflammatory cytokines and chemokines. In fact, recent evidence suggests that minocycline may attenuate the neuroinflammatory effects of opioids while enhancing their antinociceptive effects. Therefore, the investigators will determine if minocycline will mitigate OIH in methadone-maintained patients.

DETAILED DESCRIPTION:
Sixty completers will be recruited through the VA methadone clinic, as well as through the APT Foundation Methadone Maintenance Program. After the initial phone screening, potential subjects will undergo a comprehensive evaluation which will include medical, psychiatric, and drug use histories as well as physical, psychiatric, and laboratory examinations. Laboratory examination will include CBC, liver and thyroid function tests, serum electrolytes, BUN, creatinine, PT, PTT, urine analysis (including urine pregnancy for women) and urine toxicology screening.

Participants will be terminated from the study following opioid relapse, or use of any other psychotropic medications. If participants are noncompliant (no-show, positive urine screening, noncompliance with medication protocol/missing more than one dose of minocycline/placebo), participation will be terminated.

This double-blind, randomized clinical trial will randomize male and female veterans and non-veterans currently undergoing methadone maintenance treatment for opioid dependence to either minocycline (200mg/day) or placebo for 15 days. Upon inclusion, participants will be subjected to a pain assessment to evaluate baseline pain thresholds and tolerance: the Cold Pressor Test. An experimental treatment of either minocycline or placebo will then be initiated and maintained for 15 days. Additionally, at the beginning of Week 2 of treatment, participants will be given a Personal Digital Assistant (PDA) an HP iPAQ Pocket PC 2003 Pro that will administer Ecological Momentary Assessments (EMA). Using EMA, we can assess change in pain sensitivity, withdrawal symptoms and cognitive performance in the participants' natural environment, which increases the ecological validity of the study. Participants will be asked to return to the laboratory several times a week for the 15 consecutive days that they are taking minocycline in order to receive the study medication and to assess changes in pain thresholds and tolerance (i.e. to assess the presence, or lack thereof of hyperalgesia). Upon completion of experimental treatment, participants will be asked to return a final time to undergo pain measurement once more, to assess any changes in pain sensitivity after completion of minocycline.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, between the ages of 18 and 55
* Diagnosed with opioid dependence and currently enrolled in methadone maintenance treatment
* Compliant in methadone maintenance treatment and on a stable dose for two weeks or greater
* No current dependence or abuse of any other drugs (other than tobacco or marijuana)
* No current medical problems
* For women:

  * not pregnant as determined by pregnancy screening;
  * not breast feeding; u
  * using acceptable birth control methods;
  * not experiencing moderate to severe premenstrual symptoms (may interfere with pain assessment);
  * regular menstrual cycles

Exclusion Criteria:

* Current major psychiatric illnesses including mood, psychotic, or anxiety disorders
* History of major medical illnesses, including liver diseases, heart disease, or other medical conditions that the physician investigator deems contraindicated for inclusion in the study
* Current use of over-the-counter or prescription psychoactive drugs (including regular use of NSAIDS, antidepressant, anxiolytics, antipsychotics, mood stabilizers, psychostimulants) or drugs that would be expected to have major interactions with drugs to be tested, e.g., benzodiazepines, codeine, Percocet, and other opiate drugs
* Liver function tests (ALT or AST) greater than 3x normal
* Allergy to minocycline or other tetracyclines

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- VA Hospital, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-five subjects were screened. Of those, 27 were deemed eligible and enrolled.
Period: Overall Study
Arm/Group | Minocycline | Placebo
Started | 14 | 13
Completed | 10 | 10
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (4.5) | 47.9 (10.0) | 47.2 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Subjects race and ethnicity
  Participants
    Race/Ethnicity: Black | 1 | 2 | 3
    Race/Ethnicity: White | 7 | 6 | 13
    Race/Ethnicity: Hispanic | 2 | 1 | 3
    Race/Ethnicity: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pain Threshold
Description: The Cold Pressor Test (CPT) measures pain threshold (in seconds). For this test, two water coolers filled with either warm (100.04ºF/37.8ºC) or cold water (32.9-34.7ºF/0.5-1.5ºC) are used. To begin the CPT, participants first immerse their hand into the warm-water bath for 2 min. Participants are then instructed to immerse their hand into the cold water bath and report the first time they experience pain (pain threshold). Lower scores indicate lower pain threshold. Minimum score is 0 seconds, and a maximum cut-off score of 300 seconds is used to prevent tissue damage.
Time Frame: One measurement at each of 5 weekly sessions: Baseline, Day 8, Day 15, Day 22 and at Follow-up (~Day 28)
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Minocycline: This group received 200mg minocycline 1x/day for 15 days.
- Placebo: This group received a placebo capsule 1x/day for 15 days.
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
seconds
  Baseline | 18.72 (11.25) | 24.78 (13.77)
  Day 8 (Test Day 1) | 16.16 (6.46) | 24.37 (17.57)
  Day 15 (Test Day 2) | 16.13 (5.67) | 18.46 (6.86)
  Day 22 (Test Day 3) | 16.21 (5.86) | 25.75 (15.45)
  ~Day 28 (Follow-up) | 17.59 (9.34) | 21.92 (7.93)

2. Primary Outcome: Pain Tolerance
Description: The Cold Pressor Test (CPT) measures pain threshold and pain tolerance (in seconds). For this test, two water coolers filled with either warm (100.04ºF/37.8ºC) or cold water (32.9-34.7ºF/0.5-1.5ºC) are used. To begin the CPT, participants first immerse their hand into the warm-water bath for 2 min. Participants are then instructed to immerse their hand into the cold water bath and report when the pain becomes unbearable (pain tolerance). Lower scores indicate lower pain tolerance. Minimum score is 0 seconds, and a maximum cut-off score of 300 seconds is used to prevent tissue damage.
Time Frame: One measurement at each of 5 weekly sessions: Baseline, Day 8, Day 15, Day 22 and at Follow-up (~Day 28)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
seconds
  Baseline | 40.86 (21.71) | 59.72 (30.4)
  Day 8 (Test Day 1) | 37.42 (12.76) | 52.56 (28.54)
  Day 15 (Test Day 2) | 34.41 (11.84) | 48.42 (36.62)
  Day 22 (Test Day 3) | 36.61 (20.45) | 51.52 (37.53)
  ~Day 28 (Follow-up) | 31.58 (12.56) | 43.14 (15.46)

3. Secondary Outcome: Brief Pain Inventory - Short Form: Pain Severity
Description: Brief Pain Inventory - Short Form: BPI-SF is a self-report questionnaire that assesses the impact of pain on daily function, location of pain, pain medications, and amount of pain relief in the past 24 hours or the past week. Each question is scored 0-10, and the scores are summed and then averaged to create a pain severity score. Minimum score is 0; maximum score is 10. Higher scores indicate more severely perceived pain.
Time Frame: One measurement at each of 5 weekly sessions: Baseline, Day 8, Day 15, Day 22 and at Follow-up (~Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: This group received placebo 1x/day for 15 days.
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 1.28 (1.83) | 1.10 (1.93)
  Day 8 (Test Day 1) | 0.88 (1.56) | 0.95 (1.96)
  Day 15 (Test Day 2) | 0.78 (1.27) | 1.00 (1.81)
  Day 22 (Test Day 3) | 0.80 (1.30) | 1.18 (2.66)
  ~Day 28 (Follow-up) | 1.10 (1.45) | 1.28 (2.57)

4. Secondary Outcome: Brief Pain Inventory - Short Form: Interference
Description: Brief Pain Inventory - Short Form: BPI-SF is a self-report questionnaire that assesses 7 questions each rated on a scale of 0-10, which are added and divided by 7. This average score of 7 questions gives a "pain interference with living" score, with a minimum score of 0 and a maximum score of 10.
  Higher scores indicate that pain interferes more with aspects of daily life.
Time Frame: One measurement at each of 5 weekly sessions: Baseline, Day 8, Day 15, Day 22 and at Follow-up (~Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 0.93 (1.74) | 0.97 (2.37)
  Day 8 (Test Day 1) | 0.90 (1.69) | 1.33 (2.07)
  Day 15 (Test Day 2) | 0.63 (1.23) | 1.04 (2.15)
  Day 22 (Test Day 3) | 0.67 (1.30) | 1.49 (2.57)
  ~Day 28 (Follow-up) | 0.52 (0.89) | 1.2 (2.57)

5. Secondary Outcome: Opioid Withdrawal Symptom Checklist (OWSC): Back Pain Item
Description: For safety reasons, withdrawal signs and symptoms were assessed using a 22-item withdrawal instrument that has been reliably used to assess opiate withdrawal. As an additional assessment of daily pain, the presence of "back pain" item was analyzed. This item has a minimum score of 0 and maximum score of 4, with higher scores indicates more agreement with statement/more back pain.
Time Frame: One measurement at each of 5 weekly sessions: Baseline, Day 8, Day 15, Day 22 and at Follow-up (~Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 0 (0) | 0.10 (0.32)
  Day 8 (Test Day 1) | 0 (0) | 0.10 (0.7)
  Day 15 (Test Day 2) | 0.10 (0.32) | 0.20 (0.63)
  Day 22 (Test Day 3) | 0.20 (0.42) | 0.20 (0.63)
  ~Day 28 (Follow-up) | 0.10 (0.32) | 0.40 (0.97)

6. Secondary Outcome: Profile of Mood States (POMS) Depression Subscale
Description: The POMS is a 65-item scale that divides items amongst eight mood states (tension, depression, anger, fatigue, confusion, vigor) on a 5-point rating scale (0=not at all to 5=extremely). We analyzed the 15-item "Depression" subscale, which has a minimum score of 0 and a maximum score of 75. Higher score indicate more agreement with the statement/more feelings of depression.
Time Frame: One measurement at each of 5 weekly sessions: Baseline, Day 8, Day 15, Day 22 and at Follow-up (~Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 20.80 (5.33) | 18.9 (5.22)
  Day 8 (Test Day 1) | 18.9 (5.22) | 17.9 (3.35)
  Day 15 (Test Day 2) | 21.00 (6.46) | 16.7 (3.71)
  Day 22 (Test Day 3) | 19.2 (5.43) | 17.0 (5.01)
  ~Day 28 (Follow-up) | 18.8 (7.57) | 17.8 (7.87)

7. Secondary Outcome: Profile of Mood States (POMS) - Total Mood Disturbance
Description: The POMS is a 65-item scale that divides items amongst eight mood states (tension, depression, anger, fatigue, confusion, vigor) on a 5-point rating scale (0=not at all to 5=extremely). Total Mood Disturbance is calculated by adding the "tension, depression, anger, fatigue, and confusion" subscale scores and subtracting the "vigor" subscale score. This has a minimum of 0 and a maximum score of 210. Higher score indicate more mood disturbance.
Time Frame: One measurement at each of 5 weekly sessions: Baseline, Day 8, Day 15, Day 22 and at Follow-up (~Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: This group received placebo capsules 1x/day for 15 days.
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 43.1 (15.04) | 47.4 (22.63)
  Day 8 (Test Day 1) | 44.7 (14.43) | 41.88 (13.62)
  Day 15 (Test Day 2) | 50.3 (18.29) | 40.4 (15.38)
  Day 22 (Test Day 3) | 43.4 (17.51) | 42.3 (17.51)
  ~Day 28 (Follow-up) | 40.7 (15.52) | 42.2 (23.61)

8. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ): Sensory Subscale
Description: This measure is a subscale of the SF-MPQ, comprised of 11 of the 15 total items. The measure is completed immediately after the CPT, where participants describe their experience of CPT pain by choosing among a series of possible answers [none (score=0), mild (score=1), moderate (score=2), or severe (score=3)]. The items to describe the pain are 'Throbbing','Shooting', 'Stabbing', 'Sharp', 'Cramping', 'Gnawing', 'Hot/burning', 'Aching', 'Heavy', 'Tender', and 'Splitting'. The scores for these 11 items are summed as a measure of Sensory pain, with a minimum score of 0 and a maximum score of 33.
Time Frame: One measurement at each of 5 weekly sessions: Baseline, Day 8, Day 15, Day 22 and at Follow-up (~Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 10.33 (7.88) | 12.9 (8.69)
  Day 8 (Test Day 1) | 10.9 (8.32) | 13.1 (4.77)
  Day 15 (Test Day 2) | 10.8 (7.54) | 14.2 (11.05)
  Day 22 (Test Day 3) | 11.3 (8.26) | 13.3 (9.44)
  ~Day 28 (Follow-up) | 12.5 (7.8) | 10.7 (8.82)

9. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ): Affective Subscale
Description: This measure is a subscale of the SF-MPQ, comprised of 4 of the 15 total items. The measure is completed immediately after the CPT, where participants describe their experience of CPT pain by choosing among a series of possible answers [none (score=0), mild (score=1), moderate (score=2), or severe (score=3)]. The items to describe the pain are 'Tiring-Exhausting', 'Sickening', 'Fearful', 'Punishing-Cruel'. The scores for these 4 items are summed as a measure of Affective pain, with a minimum score of 0 and a maximum score of 12.
Time Frame: One measurement at each of 5 weekly sessions: Baseline, Day 8, Day 15, Day 22 and at Follow-up (~Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 2.0 (3.32) | 1.5 (2.22)
  Day 8 (Test Day 1) | 1.7 (2.11) | 1.7 (2.11)
  Day 15 (Test Day 2) | 1.9 (3.45) | 2.2 (3.74)
  Day 22 (Test Day 3) | 2.4 (3.24) | 2.0 (3.74)
  ~Day 28 (Follow-up) | 1.89 (3.48) | 2.3 (4.22)

10. Secondary Outcome: Interleukin-1 Beta (IL-1β)
Description: Serum cytokine analysis assayed using electrochemiluminescence multi-array technology (Meso Scale Discovery, Gaithersburg, MD). IL-1β is measured in pictograms per milliliter (pg/ml). Cytokines were assessed at screening (approximately 1 week prior to medication), and on the last day of medication treatment. Higher numbers indicate higher blood levels of this cytokine.
Time Frame: Pre/post : At Screening before medication, and on Day 22 of medication
Measure: Mean (Standard Deviation); unit: pictograms per milliliter
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
pictograms per milliliter
  Screening | 0.80 (0.58) | 0.72 (0.55)
  Day 22 | 0.67 (0.44) | 0.62 (0.53)

11. Secondary Outcome: Interleukin-6 (IL-6)
Description: Serum cytokine analysis assayed using electrochemiluminescence multi-array technology (Meso Scale Discovery, Gaithersburg, MD). IL-6 is measured in pictograms per milliliter (pg/ml).Cytokines were assessed at screening (approximately 1 week prior to medication), and on the last day of medication treatment. Higher numbers indicate higher blood levels of this cytokine.
Time Frame: Pre/post : At Screening before medication, and on Day 22 of medication
Measure: Mean (Standard Deviation); unit: pictograms per milliliter
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
pictograms per milliliter
  Screening | 1.64 (1.30) | 1.11 (0.94)
  Day 22 | 2.14 (1.63) | 1.99 (2.53)

12. Secondary Outcome: Tumor Necrosis Factor Alpha (TNF-α)
Description: Serum cytokine analysis assayed using electrochemiluminescence multi-array technology (Meso Scale Discovery, Gaithersburg, MD). TNF-α is measured in pictograms per milliliter (pg/ml).Cytokines were assessed at screening (approximately 1 week prior to medication), and on the last day of medication treatment. Higher numbers indicate higher blood levels of this cytokine.
Time Frame: Pre/post : At Screening before medication, and on Day 22 of medication
Measure: Mean (Standard Deviation); unit: pictograms per milliliter
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
pictograms per milliliter
  Screening | 2.86 (1.79) | 2.66 (0.80)
  Day 22 | 2.66 (0.80) | 2.53 (0.96)

13. Secondary Outcome: Ecological Momentary Assessments (EMA) - Pain
Description: Participants will be asked "Do you feel any pain at this moment" on seven-point Likert scales (1=strongly disagree to 7=strongly agree) 4 times per day outside of the laboratory (in their natural environment) using a personal digital assistant on days 8-14 of medication treatment. All scores were averaged to compute one score. Higher scores indicate more feelings of pain.
Time Frame: 4x/day for one week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.22 (0.63) | 1.14 (0.49)

14. Secondary Outcome: Ecological Momentary Assessments (EMA) - Craving
Description: Participants will be asked "Are you craving heroin at this moment" on seven-point Likert scales (1=strongly disagree to 7=strongly agree) 4 times per day outside of the laboratory (in their natural environment) using a personal digital assistant on days 8-14 of medication treatment. All scores were averaged to compute one score. Higher scores indicate more craving for heroin.
Time Frame: 4x/day for one week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.04 (0.18) | 1.14 (0.49)

15. Secondary Outcome: Ecological Momentary Assessments (EMA): SOWS
Description: Self-report opioid withdrawal scale. Withdrawal symptoms are measured on a 7-point Likert scale (1=strongly disagree, 7=strongly agree). Participants complete these ratings 4 times per day on days 8-14 of medication treatment. All scores were averaged to compute one score. Higher scores indicate more withdrawal symptoms.
Time Frame: 4x/day over one week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.05 (0.24) | 1.03 (0.22)

16. Secondary Outcome: Digit Symbol Substitution Test
Description: The DSST is a test of psychomotor performance, which measures motor persistence, sustained attention, response speed and visuomotor coordination. The task is to fill in blank spaces with the symbols that are paired with the number above the blank space as fast as possible for 90 sec. The minimum score is 0 and the maximum score is 120. Higher numbers indicate better cognitive performance.
Time Frame: Baseline (Day 0), Pre- and 1-hour post-medication treatment on Test Days 8, 15 and 22, and at Follow-up (~Day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 37.11 (8.57) | 37.11 (9.05)
  Day 8 Pre-medication | 42.33 (8.12) | 40.89 (4.96)
  Day 8 Post-medication | 41.78 (6.72) | 40.89 (5.30)
  Day 15 Pre-medication | 45.67 (8.32) | 43.33 (6.96)
  Day 15 Post-medication | 43.25 (11.51) | 41.11 (7.41)
  Day 22 Pre-medication | 48.44 (13.38) | 43.00 (7.23)
  Day 22 Post-medication | 46.56 (9.19) | 40.11 (9.16)
  ~Day 28 (Follow-up) | 50.75 (8.97) | 46.67 (5.89)

17. Secondary Outcome: Sustained Attention to Response Test (SART): No-go Trials: Errors of Commission
Description: The SART is a Go No-Go task. It assesses the ability to withhold responses to an infrequently occurring target (No-Go trials). A total of 225 single digits (25 x 9 digits) are presented on a computer monitor for 250 ms each, immediately followed by a mask for 900 ms. Subjects must press a spacebar in response to every digit except the "3". Higher numbers indicate more errors of commission.
Time Frame: Baseline (Day 0), Pre- and 1-hour post-medication treatment on Test Days 8, 15 and 22, and at Follow-up (~Day 28
Measure: Mean (Standard Deviation); unit: commission errors
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
commission errors
  Baseline | 7 (6.41) | 9 (5.4)
  Day 8 Pre-medication | 5.78 (4.6) | 8.33 (6.16)
  Day 8 Post-medication | 5.75 (5.09) | 7.33 (5.27)
  Day 15 Pre-medication | 7.40 (5.76) | 7.89 (6.47)
  Day 15 Post-medication | 5.5 (5.8) | 8.7 (5.1)
  Day 22 Pre-medication | 9.3 (5.58) | 7.3 (7.67)
  Day 22 Post-medication | 5.6 (4.78) | 9.89 (7.27)
  ~Day 28 (Follow-up) | 7.00 (4.54) | 7.26 (6.88)

18. Secondary Outcome: Sustained Attention to Response Test (SART): Go Trials: Errors of Omission
Description: The SART is a Go No-Go task. It assesses the ability to withhold responses to an infrequently occurring target (No-Go trials).The SART is a Go No-Go task. It assesses the ability to withhold responses to an infrequently occurring target (No-Go trials). A total of 225 single digits (25 x 9 digits) are presented on a computer monitor for 250 ms each, immediately followed by a mask for 900 ms. Subjects must press a spacebar in response to every digit except the "3". Higher numbers indicate more errors of omission.
Time Frame: Baseline (Day 0), Pre- and 1-hour post-medication treatment on Test Days 8, 15 and 22, and at Follow-up (~Day 28
Measure: Mean (Standard Deviation); unit: ommission errors
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 10
ommission errors
  Baseline | 10.9 (8.17) | 17.9 (16.78)
  Day 8 Pre-medication | 9.11 (12.67) | 13.78 (9.93)
  Day 8 Post-medication | 6.88 (8.08) | 13.44 (9.94)
  Day 15 Pre-medication | 15.8 (29.67) | 21 (23.81)
  Day 15 Post-medication | 7.7 (12.14) | 27 (27.87)
  Day 22 Pre-medication | 18.4 (18.71) | 25.4 (30.16)
  Day 22 Post-medication | 13.2 (12.22) | 22.33 (24.79)
  ~Day 28 (Follow-up) | 11.1 (7.69) | 21.1 (21.13)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT02359006/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT02359006/SAP_001.pdf